CLINICAL TRIAL: NCT05530200
Title: Phase II Multi-center Clinical Study of PD-1 Inhibitor Combined With Hypofractionated Radiotherapy and GM-CSF With IL-2(PRaG2.0 Regimens) Rechallenge for Patients With Resistance to PD1/PD-L1 Inhibitors in Refractory Advanced Solid Tumors.
Brief Title: PRaG Regimens Rechallenge for Patients With Resistance to PD1/PD-L1 Inhibitors in Refractory Advanced Solid Tumors.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JD-LK-2022-102-01
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiation Dose Hypofractionation; Immune Checkpoint Inhibitors; Granulocyte-Macrophage Colony-Stimulating Factor; Interleukin-2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy, PD-L1 inhibitors Sequential GM-CSF and IL-2 (Experimental)
  Interventions: Radiation: Hypofractionated radiotherapy; Drug: PD-L1 inhibitor; Drug: GM-CSF; Drug: IL-2

INTERVENTIONS:
Radiation: Hypofractionated radiotherapy — 24Gy/8Gy/3f
Drug: PD-L1 inhibitor — q3w
Drug: GM-CSF — 200μg, D1-D7
Drug: IL-2 — at a dose of 2 million IU, D8-D14

SUMMARY:
Finding an effective treatment to rescue with resistance of PD-1/PD-L1 inhibitor has been an urgent problem.The PRaG trial as a salvage therapy in advanced solid tumors has obtained satisfactory results.We found that patients with PD-1/PD-L1 inhibitors resistance are more likely to benefit from the PRaG regimens(PD-1 inhibitors combined with radiotherapy and GM-CSF with IL-2). Further phase II clinical trial was conducted to confirm the efficacy and safety of PRaG regimen rechallenge for patients with resistance to PD1/PD-L1 inhibitors in refractory advanced solid tumors.

DETAILED DESCRIPTION:
Patinets with PD-1/PD-L1 inhibitors resistance have limited treatment.ICIs rechallenge is one of the attractive and challenging selection strategies.The efficacy and safety of PD-1/PD-L1 inhibitor rechallenge remain unclear.PRaG regimens realize the sensitization of the efficacy of PD-1 inhibitors, broaden the anti-cancer spectrum of PD-1 immunotherapy, and achieve precise and minimally invasive tumor treatment.PRaG regimens might benefit the survival of patients with resistance to PD1/PD-L1 inhibitors in refractory advanced solid tumors.A phase II clinical study is planned to explore the efficacy and safety of PRaG regimens in advanced refractory solid malignancies after resistance of PD-1/PD-L1 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged≥18 years;
2. The patients must conform to the advanced solid cancer with multiple metastases(may be accompanied by metastasis of other organs),progression after first-line systemic therapy and have clear pathological diagnosis report;
3. Disease progression after PD-1/PD-L1 therapy in the past, except for the permanent discontinuation of the drug due to immune-related toxicity of grade 3 or above;
4. Enrolled patients must improve the detection of PD-L1, TMB, MSI and other immune-related indicators;
5. No congestive heart failure, unstable angina pectoris, unstable arrhythmia within the past 6 months;
6. Eastern Cooperative Oncology Group (ECOG) Performance Status: 0-3, and life expectancy 3 months or more;
7. There was no history of serious hematopoietic function, abnormal heart, lung, liver, kidney function and immune deficiency;
8. One week before enrollment,absolute value of T lymphocytes≥0.5 times of normal lower limit,neutrophil ≥ 1.0×109/L,AST and ALT ≤3.0 times normal upper limit(Liver cancer/liver metastasis patients ≤5.0 times normal upper limit),creatinine ≤ 3.0 times normal upper limit,serum calcium≥2.0mmol/L;
9. Patients must have the ability to understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with a history of other malignant diseases in the last 2 years,except cured skin cancer and carcinoma in situ;
3. Patients with a history of uncontrolled epilepsy, central nervous system diseases or mental disorders, whose clinical severity may hinder the signing of informed consent or affect the patient's compliance with drug treatment as judged by the investigator;
4. Clinically significant (ie, active) heart disease, such as symptomatic coronary heart disease, congestive heart failure New York Heart Association (NYHA) Class II or greater, or severe arrhythmia requiring drug intervention, or a history of myocardial infarction within the last 12 months;
5. Organ transplantation requiring immunosuppressive therapy;
6. Known active infection, or significant hematological, renal, metabolic,gastrointestinal, endocrine function or metabolic disorders, or other serious uncontrolled concomitant diseases as judged by the investigator;
7. Hypersensitivity to any component of the study drug;
8. History of immunodeficiency, including positive HIV test or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation, or other related diseases requiring long-term oral hormone therapy (greater than 10 mg/d prednisone);
9. Patients who are in the period of acute and chronic tuberculosis infection(patients with positive T-spot test and suspicious tuberculosis lesions on chest radiography), are in the period of acute hepatitis infection or have chronic hepatitis B virus copy number higher than the normal range;
10. Other conditions considered unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 3 years
  objective response rate

SECONDARY OUTCOMES:
PFS | Up to 3 years
  progression-free survival
DCR | Up to 3 years
  CR+PR+SD(RECIST 1.1)
OS | Up to 3 years
  overall survival
Treatment Related Severe Adverse Effects | Up to 3 years
  Number of participants with treatment-related severe adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

IPD SHARING:
Plan to Share IPD: No